CLINICAL TRIAL: NCT03736421
Title: Observational Study to Evaluate Peripheral IntraVenous Analysis (PIVA) in Euvolemic, Hypovolemic, and Hypervolemic Emergency Department Patients
Acronym: PIVA
Status: Terminated | Type: Observational
Why Stopped: Enrollment and other trial activities have temporarily paused due to COVID-19 and are expected to resume in the future; This is not a suspension of IRB approval
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Nathan Shapiro, Associate Professor of Emergency Medicine, Beth Israel Deaconess Medical Center
Other Study IDs: 2018P000494
Record Dates: First submitted 2018-10-29; First posted 2018-11-09 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Infection; Hypervolemia; Hypovolemia; Septic Shock; Acute Heart Failure; Congestive Heart Failure
MeSH Terms: conditions — Infections; Edema; Hypovolemia; Shock, Septic; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control Cohort: This cohort is recruited to help to define what a "normal" PIVA value should be during a state of presumed euvolemia.
  Interventions: Procedure: Peripheral Intravenous Analysis (PIVA); Diagnostic Test: Passive leg raise (PLR)
- Infection Cohort: This cohort are subjects with suspected infection, enriched to contain sepsis patients.
  Interventions: Procedure: Peripheral Intravenous Analysis (PIVA); Procedure: Non-invasive fluid response measure; Diagnostic Test: Passive leg raise (PLR)
- Acute Heart Failure: This cohort will have a diagnosis of CFH who are being admitted to the hospital. These patients will be followed during their hospital course.
  Interventions: Procedure: Peripheral Intravenous Analysis (PIVA); Procedure: Non-invasive fluid response measure; Diagnostic Test: Passive leg raise (PLR)

INTERVENTIONS:
Procedure: Peripheral Intravenous Analysis (PIVA) — Non-invasive measurement of peripheral intravenous waveform analysis (PIVA) obtained by connecting an Edwards standard transducer to a universal adaptor or stopcock on a peripheral IV
  Other Names: PIVA
Procedure: Non-invasive fluid response measure — To measure the stroke volume and changes in stroke volume in response to a passive leg raise (PLR) maneuver and fluid administration.
  Groups: Acute Heart Failure; Infection Cohort
Diagnostic Test: Passive leg raise (PLR) — Test to predict cardiac output and fluid responsiveness
  Other Names: PLR

SUMMARY:
The overall goal of this multicenter project is to characterize the expected normal range of Peripheral IntraVenous Volume Analysis (PIVA) values during a euvolemic state, and how those ranges may be altered by comorbidities; the relationship between PIVA and intravenous volume administration during resuscitation of infected patients with presumed hypovolemia; and, the relationship between PIVA and volume decreases during diuresis in acute heart failure patients with hypervolemia.

DETAILED DESCRIPTION:
The determination of volume status remains a clinical challenge in medicine. Patients may develop hypovolemia (too little fluids in the vascular space) due to conditions such as hemorrhage, dehydration, or infection with vascular leak. Alternatively, patients may become hypervolemic (too much fluids in the vascular space), due to conditions such as heart failure, renal failure, or iatragenic over-resuscitation all of which overwhelm the kidney's ability to regulate intravascular volume status. In clinical practice, clinicians strive to return patients to euvolemia (the "right" volume status) through the administration of intravenous fluids or diuretics which remove fluids to achieve homeostasis. While there are a number of proposed clinical exam findings (e.g. dry mucous membranes or skin turgor), measurements (e.g. central venous pressure), or laboratory tests (e.g. blood urea nitrogen), none are precise or universally accepted as reliable methodologies to assess volume status.

The goal of this study is to perform a prospective observational study on three distinct cohorts during ED presentation to assess the variability and performance of PIVA in tracking volume status.

ELIGIBILITY:
Control Cohort (Presumed Euvolemia)

Inclusion Criteria:

* Age > 18 years old
* Assessed as "euvolemic" by treating physician

Exclusion Criteria:

* History of any type of decreased oral intake or volume loss (e.g. diarrhea, vomiting, etc)
* History of a fever
* History of bleeding
* Any acute illness expected to alter volume
* Known or suspected pregnancy
* Active irregular heart rhythm
* In the opinion of the treating physician, no anticipated intravenous fluid administration
* History of chronic or end stage renal disease
* Liver failure
* History of Acute heart failure
* Presence of abnormal vital signs (90 < HR < 60; 180 < SBP < 110, respiratory rate > 20, pulse ox < 92% or need for supplemental oxygen, 99.0 < temperature < 96).

  2 additional group will be included in this euvolemic group
* Non-elderly patients (age < 50 year) without any comorbid illnesses and
* Age >65
* Diabetes on medications
* Hypertension on medications
* Vascular disease defined by history of peripheral vascular disease, stroke, MI

Note: patients that receive >250 cc of IVF will be excluded from analysis.

Infection Cohort (Presumed Hypovolemia)

Inclusion Criteria:

* Age > 18 years old
* An accessible intravenous catheter is in place
* Known or suspected infection as assessed by the clinical team
* Intention to admit to the hospital
* Anticipated administration of intravenous fluids per clinical team

Exclusion Criteria:

* Clinical exam consistent with volume overload
* Known or suspected pregnancy
* Patients with a history of chronic renal insufficiency or end-stage renal disease
* Patients with a history of acute heart failure

Acute Heart Failure (Hypervolemic cohort)

Inclusion Criteria:

* Age > 17 years old
* An accessible intravenous catheter is in place
* Primary clinical diagnosis of CHF
* Meet 2 of the three criterion:
* X-ray diagnosis
* Elevated bnp from known baseline
* Clinical diagnosis
* Received or intent to administer a diuretic agent
* Intent to admit to the hospital for anticipated > 24 hour period

Exclusion Criteria:

* History of any type of decreased oral intake or volume loss (e.g. diarrhea, vomiting, etc)
* History of a fever
* History of bleeding
* Known or suspected pregnancy
* Active irregular heart rhythm
* History of dialysis dependent end stage renal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Presumed Euvolemia cohort: This cohort is recruited to help to define what a "normal" PIVA value should be during a state of presumed euvolemia.
  Presumed Hypovolemia cohort: This is a cohort of patients with suspected infection and enriched with categories of sepsis patients.
  Hypervolemic cohort: This is a cohort of patients with a diagnosis of Congestive Heart Failure (CHF) who are being admitted to the hospital.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-11-10 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Association between PIVA measurement and fluid status (net gain vs net loss) | Baseline to 6 hours for euvolemic and hypovolemic cohort, and baseline to 72 hours for hypervolemic cohort
  Change in fluid status over the first 6 hours as measured by weight and urine output and pressure status from the Edwards transducer

SECONDARY OUTCOMES:
Response to Passive leg raise | For the euvolemic cohort, baseline to 2 hours; For hypovolemic, cohort baseline to 6 hours; for the hypervolemic cohort, baseline up to 72 hours
  Compute the change in PIVA measurement between before and after the passive leg raise challenge within each cohort
Association between PIVA and non-invasive monitoring responsiveness to passive leg raise | Baseline up to 72 hours
  Compare change in PIVA measurements to non-invasive monitoring measurements before and after passive leg raise and before and after fluid boluses

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Beth Israel Medical Center, Boston, Massachusetts
  - St. Vincent Hospital, Worcester, Massachusetts
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No